CLINICAL TRIAL: NCT07334613
Title: The Impact of Alienation on the Psychological and Social Aspects and Quality of Life of Medical Students in Assuit University
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Khaled Mohamed Mohamed, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: alienation on the psychologica
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Alienation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: the international ,and those from other governorates, medical students in faculty of medicine in assuit university

SUMMARY:
________________________________________ Medical education is one of the most challenging and demanding academic paths, often associated with high levels of stress, workload, and continuous pressure to achieve academic excellence [1,2,4,5]. These factors can significantly affect the psychological and social well-being of medical students, especially during their formative years at university [6,7].

One of the critical psychological phenomena that may emerge in this context is alienation, which refers to a sense of estrangement, disconnection, or detachment from oneself, others, or the surrounding environment [3,8]. Alienation among medical students has been linked to various psychological consequences, including anxiety, depression, burnout, and a reduced sense of personal accomplishment [4-7,11-13].

On a social level, alienation can hinder the development of healthy interpersonal relationships, reduce social participation, and impair the sense of belonging within the academic community [8-10,13,15]. These psychological and social challenges, in turn, can have a profound impact on students' overall quality of life, which encompasses their physical, emotional, and social well-being [10,14].

Understanding the impact of alienation on medical students is of particular importance in contexts such as Assiut University, where cultural, social, and academic pressures may further intensify the experience of alienation [11-13]. Investigating this relationship can help educators, administrators, and policymakers develop targeted interventions and supportive strategies that promote students' psychological health, social integration, and overall academic success [9,10,13,15].

This study, therefore, aims to explore the impact of alienation on the psychological and social aspects of medical students at Assiut University, and how these factors collectively influence their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* international students of faculty of medicine in assuit university.
* students from governorates other than assuit.

Exclusion Criteria:

* cases with psychiatric disorder prior to study.
* cases with any physical or medical disease.
* refusal of cases to participate in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: international students of faculty of medicine in assuit university and students from governorates other than assuit.
Sampling Method: Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
assessmet of quality of life in foreigner students | baseline
  WHO Quality of Life (WHOQOL) is an internationally validated instrument developed by the World Health Organization to assess individuals' perceptions of their position in life within the context of culture, value systems, personal goals, expectations, and concerns. It covers domains such as physical health, psychological well-being, social relationships, and environment (WHOQOL Group, 1998).